CLINICAL TRIAL: NCT06273371
Title: Tolerance and Growth Outcomes in Children Diagnosed With Cow's Milk Protein Allergy and Prescribed an Extensively Hydrolyzed Casein Formula (Damira 2000©) in Spain
Acronym: DELISA
Status: Completed | Type: Observational
Sponsor: Lactalis (Industry)
Responsible Party: Sponsor
Other Study IDs: DELISA2023
Record Dates: First submitted 2024-02-06; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cow's Milk Protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Damira 2000 Infant formula — 100% extensive casein hydrolysate Infant formula

SUMMARY:
Damira 2000© is a 100% extensive casein hydrolysate (eHCF). It is formulated to help reverse growth retardation as a result of cow's milk proteins allergy (CMPA), to be well tolerated and to help improve symptoms.Damira 2000 is indicated for allergy/intolerance to cow's milk proteins, atopic dermatitis secondary to CMPA, intestinal malabsorption processes and prevention of allergy/intolerance to cow's milk proteins.The study aimed at evaluating the tolerance of Damira 2000 in a cohort of children with CMPA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of allergy to cow's milk protein (CMPA): either confirmed through a placebo-controlled food challenge (DBPCFC) or highly suspected based on specific suggestive symptoms;
2. Patients under the age of 1 year at the time of cow's milk protein allergy diagnosis.
3. Patients taken Damira 2000 for at least 4 months at the time of data extraction.
4. Patients with information available on child growth (weight and height) and the following anthropometric indices at diagnosis and for at least 2 follow-up visits after first hospital visit/4 months*: Z-scores for weight-for-age (WAZ), height-for-age (HAZ), weight-for-height (WHZ) and body mass index (BMI)-for-age (BAZ).

Exclusion Criteria:

1. Patients who used other infant formulae or breast milk in addition to the study product of interest during the retrospective study period.
2. Premature children with a low birth-weight (<2.5 kg).
3. Patients diagnosed with a metabolic condition that impacts development and growth.
4. Patients diagnosed with a congenital condition and/or with prior or current disease that in the opinion of the investigator could potentially interfere with the aim of the study.

Ages: 0 Months to 12 Months | Sex: All
Age Groups: Child
Study Population: Infants aged from 0 to 12 months with cow's milk protein allergy
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Tolerance | Day 0 : V0 First visit to the hospital
  The good tolerance of the currently on the market Damira 2000 formula will be evaluated by the number and percentage of patients with no (=0) immediate allergic reactions or intestinal reactions.
  Immediate reactions are defined as those allergic reactions occurring within 1 hour after intake.
  Intestinal reactions: delayed reactions (develop after ≥ 2 hours of consumption) involving gastrointestinal (GI) tract.

SECONDARY OUTCOMES:
Weight | V1, V2 (4 months)
  To evaluate the effect of Damira 2000 on growth outcomes using weight and the related Z-scores weight-for-age (WAZ)
Height | V1, V2 (4 months)
  To evaluate the effect of Damira 2000 on growth outcomes using height and the related Z-scores height-for-age (HAZ).
Weight for height and BMI | V1, V2, (4 months)
  To evaluate the effect of Damira 2000 on growth outcomes using height and weight to calculate the Z-score weight-for-height (WHZ) and BMI for age (BAZ).
Head circumference | V1, V2 (4 months)
  To evaluate the effect of Damira 2000 on growth outcomes using Head circumference and the related Z-Score Head circumference for age.

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Quirónsalud de Córdoba, Córdoba, Andalusia
  - H. Virgen del Rocío, Seville, Andalusia
  - H. Virgen Macarena, Seville, Andalusia
  - Instituto Hispalense de pediatría, Seville, Andalusia
  - Hospital Materno infantil de Ourense, Ourense, Galicia
  - H. Clínico de Santiago, Santiago de Compostela, Galicia
  - Clínica privada Dr. Romera, Madrid
  - Fundación Jiménez Día, Madrid

IPD SHARING:
Plan to Share IPD: No